CLINICAL TRIAL: NCT03975868
Title: Risk Factors for Cut-out After Internal Fixation of Trochanteric Fractures in Elderly Subjects.
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 30342858
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Proximal Femoral Fracture
Keywords: Cut-out; Gamma nail; Lag-screw; Tip-apex distance; Trochanteric fracture
MeSH Terms: conditions — Proximal Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of associated factors for cut-out in internal fixation of extracapsular proximal femoral fracture. — Identification of factors for mechanical failure of internal fixation of extracapsular proximal femoral fracture in over 75 year olds

SUMMARY:
Proximal femoral fracture is associated with severe morbidity and mortality and high socioeconomic costs. The main mechanical complication of internal fixation in trochanteric fracture is lag-screw cut-out through the femoral head. Several factors are involved, but remain controversial. The aim of the present study was to determine risk factors for cut-out in internal fixation of extracapsular proximal femoral fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years of age
* Operated on for extracapsular proximal femoral fracture
* After bodyheight fall

Exclusion Criteria:

* Intra-capsular fractures
* trochantero-diaphyseal fractures
* subtrochanteric fractures
* fractures involving pathological bone

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 years old operated on for extracapsular proximal femoral fracture.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Mechanical failure defined by varus fracture collapse and lag-screw cut-out with extrusion through the femoral head | 3 months

IPD SHARING:
Plan to Share IPD: No